CLINICAL TRIAL: NCT05792566
Title: Development and Usability Testing of the ATOMIC Mobile App to Increase Physical Activity (PA) Levels in Children, Adolescent and Young Adults (AYA) Survivors of Childhood Cancer
Brief Title: ATOMIC Mobile App to Increase Physical Activity (PA) Levels in Survivors of Childhood Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Connecticut Children's Medical Center (Other)
Collaborators: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Tiffany Ruiz, Principal Investigator, Connecticut Children's Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-156
Record Dates: First submitted 2023-03-10; First posted 2023-03-31 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Pediatric Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: There are 3 phases of this study:
  1. Participants will be shown features from the ATOMIC app and asked to discuss what features they like and what additional content, features and functionalities they would want for a specific PA app focused on pediatric cancer survivors. This information will be used to adapt the app.
  2. Use a "talking aloud" approach as they encounter issues with completing a series of tasks related to using the app. The design team and the research team will develop a new iteration of the platform that will then be vetted by our app creation committee and the next interview participants.
  3. "Real Life" Usability Testing. 6 pediatric cancer survivors. Individualized aerobic and resistance exercise intervention. The social-cognitive-theory-based mobile app will support the exercise intervention. One-on-one messaging chats with a PA coach through the mobile app will facilitate exercise goal establishment and attainment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Real life usability testing (Experimental): B) "Real Life" Usability Testing. We will conduct a "real life" usability test in a sample of 6 pediatric cancer survivors. EX@HOME: Patients will perform an individualized aerobic and resistance exercise intervention, choosing from a list of PA, progressing from light to moderate-to-vigorous intensity totaling 30-45 min/d, 4-5 weekly/wk. for 4 weeks. The social-cognitive-theory-based mobile app will support the exercise intervention. One-on-one messaging chats with a PA coach through the mobile app will facilitate exercise goal establishment and attainment.
  Interventions: Other: Atomic app

INTERVENTIONS:
Other: Atomic app — Using the Atomic app to improve physical activity

SUMMARY:
Development and Usability Testing of the ATOMIC Mobile App to Increase Physical Activity (PA) Levels in Children, Adolescent and Young Adults (AYA) survivors of childhood cancer

DETAILED DESCRIPTION:
The purpose of this program of research is to (1) determine the adaptations required of a pre-existing mobile fitness app to tailor it for childhood cancer survivors using a behavioral theory driven approach (Social Cognitive Theory) and (2) develop and evaluate the usability of the adapted mobile app using the Technology Assessment Model. The Technology Assessment Model (TAM), which theorizes the individuals' intentions to use information technology, is based on two driving factors: perceived usefulness and perceived ease of use. Future studies will evaluate the feasibility and effectiveness of this app.

ELIGIBILITY:
Inclusion Criteria:

* Children, adolescent and young adults (AYA) ages 10 to 30 years
* diagnosis with a pediatric cancer diagnosis that requires the treatment of anthracycline therapy
* Able to speak English fluently (App currently only in English at this time)

Exclusion Criteria:

* Pediatric cancer survivors who will not be treated with anthracycline therapy
* Unable to cooperate with interviewing
* Unable to understand the content of interviews
* Non-English speaking

Ages: 10 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2023-06-12 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Ease of use and user errors will be documented for each individual during usability testing, by completing several tasks while navigating the mobile app platform | 1 year
  The interviewers will record how well the participants are able to navigate the task by recording either "easy to find", "with prompting", or "unable to complete", representing completing the task completely on their own, with help from the interviewer, or unable to complete after prompting from the interviewer. The frequency of user errors will be calculated.
The Acceptability E-Scale is six-item tool that has been validated for assessing the usability, acceptability, and satisfaction of web based programs with statements ranked on a five point scale from very difficult to very easy | 1 year
  Acceptability of a program has been proposed to be represented by obtaining a score of 24 or more.81 Good internal consistency (alpha = 0.76) as well as good initial validity has been reported. The acceptability E-scale will be administered at the completion of the "in laboratory" testing and "real-life" usability testing.

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany L Berthod (Ruiz), MSN, Principal Investigator — CT Children's Medical Center
Locations (1):
- Connecticut Children's Medical Center, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No